CLINICAL TRIAL: NCT00659828
Title: Effects of Leptin Replacement in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Richard Bookman, Associate Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20060295; 2R01DK058851-03 (NIH)
Record Dates: First submitted 2008-04-09; First posted 2008-04-16 (Estimated); Results first posted 2020-02-13 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Obesity; Metabolic Syndrome; Diabetes
Keywords: Congenital leptin deficiency; Obesity; Metabolic Syndrome; Diabetes
MeSH Terms: conditions — Obesity; Metabolic Syndrome; Diabetes Mellitus | interventions — recombinant methionyl human leptin; metreleptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Recombinant Methionyl Human Leptin (Experimental): Recombinant methionyl human leptin: Recombinant methionyl human leptin, subcutaneous, once a day, 0.02 to 0.04 mg/kg (adjusted according to weight loss).
  Interventions: Drug: Recombinant methionyl human leptin

INTERVENTIONS:
Drug: Recombinant methionyl human leptin — Recombinant methionyl human leptin, subcutaneous, once a day, 0.02 to 0.04 mg/kg (adjusted according to weight loss), indeterminate duration.
  Other Names: Metreleptin; r-metHuLeptin

SUMMARY:
To assess the endocrine and immune effects of leptin replacement in leptin-deficient children, from a consanguineous family. The hypothesis is that leptin replacement will have significant effects on endocrine function.

DETAILED DESCRIPTION:
The proposed study of the treatment of a child with congenital leptin deficiency will permit to elucidate key aspects of human endocrine function, and will give new insights on the role of leptin in human endocrine regulation.

ELIGIBILITY:
Inclusion Criteria:

* Children with a functional leptin gene mutation from a consanguineous Turkish family. Only one leptin-naïve child from this family is alive and eligible.

Exclusion Criteria:

* N/A

Ages: 5 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2005-06 (Actual); Primary Completion 2010-04-16 (Actual); Study Completion 2010-04-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julio Licinio, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Center on Pharmacogenomics, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baicy K, London ED, Monterosso J, Wong ML, Delibasi T, Sharma A, Licinio J. Leptin replacement alters brain response to food cues in genetically leptin-deficient adults. Proc Natl Acad Sci U S A. 2007 Nov 13;104(46):18276-9. doi: 10.1073/pnas.0706481104. Epub 2007 Nov 6. PMID 17986612
- [Background] Licinio J, Ribeiro L, Busnello JV, Delibasi T, Thakur S, Elashoff RM, Sharma A, Jardack PM, Depaoli AM, Wong ML. Effects of leptin replacement on macro- and micronutrient preferences. Int J Obes (Lond). 2007 Dec;31(12):1859-63. doi: 10.1038/sj.ijo.0803703. Epub 2007 Aug 7. PMID 17684509
- [Background] Licinio J, Milane M, Thakur S, Whelan F, Yildiz BO, Delibasi T, de Miranda PB, Ozata M, Bolu E, Depaoli A, Wong ML. Effects of leptin on intake of specific micro- and macronutrients in a woman with leptin gene deficiency studied off and on leptin at stable body weight. Appetite. 2007 Nov;49(3):594-9. doi: 10.1016/j.appet.2007.03.228. Epub 2007 Apr 6. PMID 17517446
- [Background] Williamson DA, Ravussin E, Wong ML, Wagner A, Dipaoli A, Caglayan S, Ozata M, Martin C, Walden H, Arnett C, Licinio J. Microanalysis of eating behavior of three leptin deficient adults treated with leptin therapy. Appetite. 2005 Aug;45(1):75-80. doi: 10.1016/j.appet.2005.01.002. PMID 15949871
- [Background] Matochik JA, London ED, Yildiz BO, Ozata M, Caglayan S, DePaoli AM, Wong ML, Licinio J. Effect of leptin replacement on brain structure in genetically leptin-deficient adults. J Clin Endocrinol Metab. 2005 May;90(5):2851-4. doi: 10.1210/jc.2004-1979. Epub 2005 Feb 15. PMID 15713712
- [Background] Licinio J, Caglayan S, Ozata M, Yildiz BO, de Miranda PB, O'Kirwan F, Whitby R, Liang L, Cohen P, Bhasin S, Krauss RM, Veldhuis JD, Wagner AJ, DePaoli AM, McCann SM, Wong ML. Phenotypic effects of leptin replacement on morbid obesity, diabetes mellitus, hypogonadism, and behavior in leptin-deficient adults. Proc Natl Acad Sci U S A. 2004 Mar 30;101(13):4531-6. doi: 10.1073/pnas.0308767101. Epub 2004 Mar 9. PMID 15070752
- [Background] Mantzoros CS, Ozata M, Negrao AB, Suchard MA, Ziotopoulou M, Caglayan S, Elashoff RM, Cogswell RJ, Negro P, Liberty V, Wong ML, Veldhuis J, Ozdemir IC, Gold PW, Flier JS, Licinio J. Synchronicity of frequently sampled thyrotropin (TSH) and leptin concentrations in healthy adults and leptin-deficient subjects: evidence for possible partial TSH regulation by leptin in humans. J Clin Endocrinol Metab. 2001 Jul;86(7):3284-91. doi: 10.1210/jcem.86.7.7644. PMID 11443202
- [Background] Ozata M, Ozdemir IC, Licinio J. Human leptin deficiency caused by a missense mutation: multiple endocrine defects, decreased sympathetic tone, and immune system dysfunction indicate new targets for leptin action, greater central than peripheral resistance to the effects of leptin, and spontaneous correction of leptin-mediated defects. J Clin Endocrinol Metab. 1999 Oct;84(10):3686-95. doi: 10.1210/jcem.84.10.5999. PMID 10523015
- [Background] Strobel A, Issad T, Camoin L, Ozata M, Strosberg AD. A leptin missense mutation associated with hypogonadism and morbid obesity. Nat Genet. 1998 Mar;18(3):213-5. doi: 10.1038/ng0398-213. No abstract available. PMID 9500540
- [Derived] Paz-Filho G, Wong ML, Licinio J. The procognitive effects of leptin in the brain and their clinical implications. Int J Clin Pract. 2010 Dec;64(13):1808-12. doi: 10.1111/j.1742-1241.2010.02536.x. PMID 21070531
- [Derived] Paz-Filho GJ, Delibasi T, Erol HK, Wong ML, Licinio J. Cellular immunity before and after leptin replacement therapy. J Pediatr Endocrinol Metab. 2009 Nov;22(11):1069-74. doi: 10.1515/jpem.2009.22.11.1069. PMID 20101893
- [Derived] Paz-Filho G, Delibasi T, Erol HK, Wong ML, Licinio J. Congenital leptin deficiency and thyroid function. Thyroid Res. 2009 Nov 4;2(1):11. doi: 10.1186/1756-6614-2-11. PMID 19889232
- [Derived] Paz-Filho GJ, Babikian T, Asarnow R, Delibasi T, Esposito K, Erol HK, Wong ML, Licinio J. Leptin replacement improves cognitive development. PLoS One. 2008 Aug 29;3(8):e3098. doi: 10.1371/journal.pone.0003098. PMID 18769731

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Recombinant Methionyl Human Leptin
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Recombinant Methionyl Human Leptin
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Weight
Time Frame: Baseline, 58 months
Measure: Number; unit: lbs
Arm/Group | Recombinant Methionyl Human Leptin
Number analyzed (Participants) | 1
lbs | NA — Results not reported due to participant confidentiality.

2. Secondary Outcome: Glucose Levels
Time Frame: Baseline, 58 months
Measure: Number; unit: mg/dL
Arm/Group | Recombinant Methionyl Human Leptin
Number analyzed (Participants) | 1
mg/dL | NA — Results not reported due to participant confidentiality.

3. Secondary Outcome: Bone Mineral Density
Time Frame: Baseline, 58 months
Measure: Number; unit: g/cm^2
Arm/Group | Recombinant Methionyl Human Leptin
Number analyzed (Participants) | 1
g/cm^2 | NA — Results not reported due to participant confidentiality.

ADVERSE EVENTS:
Time Frame: 4 years and 10 months
Description: Adverse Events not reported due to participant confidentiality.
Arm/Group | Recombinant Methionyl Human Leptin
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
This is a compassionate use study for a rare disease population. To protect participant privacy and maintain confidentiality, results will not be reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes